CLINICAL TRIAL: NCT02096653
Title: Randomized, Controlled, Double-blind, Comparative-effectiveness Study Comparing Fluoroscopically-guided and Landmark-guided Sacroiliac Joint Injections
Brief Title: Fluoroscopically-guided Versus Landmark-guided Sacroiliac Joint Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); Milton S. Hershey Medical Center (Other); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00092414
Record Dates: First submitted 2014-03-22; First posted 2014-03-26 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Sacroiliac Joint Pain
Keywords: sacroiliac joint; low back pain; steroid injection
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- X-ray guided intra-articular injection (Experimental): Injection of 40 mg depomethylprednisolone and 2 ml 0.5% bupivacaine into the SI (sacroiliac joint) cavity under fluoroscopic guidance
  Interventions: Procedure: X-ray SI joint steroid injection
- Landmark-guided SI joint injection (Active Comparator): Injection of 40 mg depomethylprednisolone and 2 ml 0.5% bupivacaine at the point of maximal tenderness (3 ml)
  Interventions: Procedure: Landmark-guided SI steroid injection

INTERVENTIONS:
Procedure: X-ray SI joint steroid injection — Injection of steroid and local anesthetic into the joint cavity using fluoroscopic guidance
  Arms: X-ray guided intra-articular injection
Procedure: Landmark-guided SI steroid injection — Injection of steroid into the joint area based on palpation. The injection may be inside the joint (intra-articular) or outside the joint in the ligaments (extra-articular)
  Arms: Landmark-guided SI joint injection

SUMMARY:
In this study, the investigators are attempting to determine whether intra- or extra-articular injections are more effective; the relative prevalence rate of intra-articular and extra-articular SI joint pain; and the accuracy of extra-articular injections using fluoroscopy as the reference standard. 124 consecutive patients with mechanical low back pain below L5, tenderness overlying the SI joint(s) and at least 3 positive provocative maneuvers will be randomized to receive SI joint injections by 2 different approaches.

Group 1 will receive fluoroscopically-guided injections into the joint. Group 2 will receive landmark-guided injections into the tender area around the joint. In order to determine whether the injection in group 2 was intra-articular or extra-articular, an x-ray will be done after the injection to ascertain the location of contrast spread. The primary outcome measure will be pain relief at 1-month. Patients who obtain benefit at 1-month will be followed at 3-months, while those who fail to obtain benefit will exit the study to receive alternative care.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18;
2. Low back pain principally below the L5 vertebra;
3. Three out of 6 positive SI joint provocative maneuvers;
4. Agreed to undergo SI joint injection for diagnostic/ therapeutic purposes;
5. Average pain score > 3/10 over the past week;
6. Pain duration > 6 weeks;

Exclusion Criteria:

1. Previous SI joint injection;
2. Leg pain > back pain or lower leg pain > upper leg pain
3. Active inflammatory spondyloarthropathy (e.g. ankylosing spondylitis);
4. Untreated coagulopathy;
5. Allergy to contrast dye or bupivacaine;
6. Pain > 20 years in duration;
7. Poorly controlled psychiatric (e.g. PTSD) or medical (congestive heart failure) condition

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Average Back Pain at 1 Month Measured Using the Numeric Pain Scale | 1 month from the start of treatment
  This outcome measure compares the average back pain at baseline to the average back pain 1 month after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The group receiving fluoroscopically-guided intra-articular injection is compared to the group receiving landmark-guided injections.

SECONDARY OUTCOMES:
Outcomes Related to Disability Measured at 1 Month Using the Oswestry Disability Index | 1 month after the start of treatment
  Functional capacity measured using Oswestry disability index. The range of possible scores for Oswestry Disability Index are 0-100. 0 is equated with no disability and 100 is the maximum disability possible.
Worst Back Pain at 1 Month Measured Using the Numeric Pain Scale | 1 month from the start of treatment
  This outcome measure compares the worst back pain at baseline to the worst back pain at 1 months after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The group receiving fluoroscopically-guided intra-articular injection is compared to the group receiving landmark-guided injections.
Average Back Pain at 3 Months Measured Using the Numeric Pain Scale | 3 months from the start of treatment
  This outcome measure compares the average back pain at baseline to the average back pain at 3 months after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The group receiving fluoroscopically-guided intra-articular injection is compared to the group receiving landmark-guided injections.
Worst Back Pain at 3 Months Measured Using the Numeric Pain Scale | 3 months after the start of treatment
  This outcome measure compares the worst back pain at baseline to the worst back pain at 3 months after the start of treatment. This is measured using the Numeric Pain Scale. The Numeric Pain Scale ranges from 0-10. 0 being no pain at all and 10 being the worst imaginable pain possible. The group receiving fluoroscopically-guided intra-articular injection is compared to the group receiving landmark-guided injections.
Outcomes Related to Disability Measured at 3 Month Using the Oswestry Disability Index | 3 months after the start of treatment
  Functional capacity measured using Oswestry disability index. The range of possible scores for Oswestry Disability Index are 0-100. 0 is equated with no disability and 100 is the maximum disability possible.
Patient satisfaction of the procedure at 1 month measured using the Likert Scale | 1 month
  Patient satisfaction is measured at 1 month after the procedure using the Likert Scale. The range of possible scores for the Likert Scale are 1-5. I being very unsatisfied and 5 being very satisfied.
Patient satisfaction of the procedure at 3 months measured using the Likert Scale | 3 months
  Patient satisfaction is measured at 1 month after the procedure using the Likert Scale. The range of possible scores for the Likert Scale are 1-5. I being very unsatisfied and 5 being very satisfied.
Positive categorical outcome | 1 month
  Decrease in average back pain score at 1 month of greater or equal to 2 points coupled with a satisfaction score > 3 on a 1-5 scale
Positive categorical outcome | 3 months
  Decrease in average back pain score at 3 months of greater or equal to 2 points coupled with a satisfaction score > 3 on a 1-5 scale
Positive diagnostic blocks | 6 hours
  The percentage of participants who experience greater or equal to 50% pain relief based on their pain diary

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Naval Hospital-San Diego, San Diego, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Rockville, Maryland
  - Penn State, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SP, Chen Y, Neufeld NJ. Sacroiliac joint pain: a comprehensive review of epidemiology, diagnosis and treatment. Expert Rev Neurother. 2013 Jan;13(1):99-116. doi: 10.1586/ern.12.148. PMID 23253394
- [Derived] Cohen SP, Bicket MC, Kurihara C, Griffith SR, Fowler IM, Jacobs MB, Liu R, Anderson White M, Verdun AJ, Hari SB, Fisher RL, Pasquina PF, Vorobeychik Y. Fluoroscopically Guided vs Landmark-Guided Sacroiliac Joint Injections: A Randomized Controlled Study. Mayo Clin Proc. 2019 Apr;94(4):628-642. doi: 10.1016/j.mayocp.2018.08.038. Epub 2019 Mar 8. PMID 30853260